CLINICAL TRIAL: NCT01451853
Title: Safety and Efficacy Study of SPI-1005 for Prevention of Chemotherapy Induced Hearing Loss
Brief Title: SPI-1005 for Prevention and Treatment of Chemotherapy Induced Hearing Loss
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sound Pharmaceuticals, Incorporated (Industry)
Collaborators: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPI-3005-201
Record Dates: First submitted 2011-10-07; First posted 2011-10-14 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Lung Cancer; Head and Neck Cancer; Hearing Loss; Ototoxicity; Tinnitus; Neuropathy
Keywords: Lung Cancer; Head and Neck Cancer; Hearing Loss; Ototoxicity; Tinnitus; Deafness; SPI-1005; Cisplatin; Carboplatin; Ebselen
MeSH Terms: conditions — Lung Neoplasms; Head and Neck Neoplasms; Hearing Loss; Ototoxicity; Tinnitus; Deafness | interventions — ebselen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SPI-1005 Low Dose (Active Comparator): 200 mg SPI-1005, capsule, po, bid, x3d surrounding each cycle of chemotherapy
  Interventions: Drug: SPI-1005 Low Dose
- SPI-1005 Middle Dose (Active Comparator): 400 mg SPI-1005, capsule, po, bid, x3d surrounding each cycle of chemotherapy
  Interventions: Drug: SPI-1005 Middle Dose
- SPI-1005 High Dose (Active Comparator): 600 mg SPI-1005, capsule, po, bid, x3d surrounding each cycle of chemotherapy
  Interventions: Drug: SPI-1005 High Dose
- Placebo (Placebo Comparator): 0 mg SPI-1005, capsule, po, bid, x3d surrounding each cycle of chemotherapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPI-1005 Low Dose — Oral capsules, 200 mg ebselen, twice daily, 3 days for each cycle of chemotherapy
  Arms: Low Dose
  Other Names:
  200 mg Ebselen
  Other Names: 200 mg Ebselen
  Arms: SPI-1005 Low Dose
Drug: SPI-1005 Middle Dose — Oral capsules, 400 mg ebselen, twice daily, 3 days for each cycle of chemotherapy
  Other Names: 400 mg Ebselen
  Arms: SPI-1005 Middle Dose
Drug: SPI-1005 High Dose — Oral capsules, 600 mg ebselen, twice daily, 3 days for each cycle of chemotherapy
  Other Names: 600 mg Ebselen
  Arms: SPI-1005 High Dose
Drug: Placebo — Oral capsules, 0 mg ebselen, twice daily, 3 days for each cycle of chemotherapy
  Other Names: 0 mg Ebselen
  Arms: Placebo

SUMMARY:
Chemotherapy treatment with platinum based agents is well noted to cause ototoxicity. It is the objective of this study to determine the safety and efficacy of SPI-1005 at three dose levels when delivered orally twice daily for 3 days, surrounding each cycle of platinum chemotherapy in head and neck or non-small cell lung cancer patients to prevent and treat chemotherapy induced hearing loss and tinnitus.

DETAILED DESCRIPTION:
Chemotherapy treatment with the platinum containing chemotherapies (e.g. cisplatin, carboplatin) are well noted and studied for their ability to cause ototoxicity which includes hearing loss, tinnitus, vertigo, or dizziness. It is the objective of this study to determine the safety and efficacy of SPI-1005 at three dose levels when delivered orally twice daily for 3 days, surrounding each cycle of platinum chemotherapy for head and neck or non-small cell lung cancer patients to prevent and treat chemotherapy induced hearing loss and tinnitus.

SPI-1005, a proprietary oral formulation of ebselen is a small molecule mimic and inducer of the enzyme Glutathione Peroxidase. GPx reduces reactive oxygen species (ROS) by reacting with glutathione. SPI-1005 has been shown to reduce cisplatin induced hearing threshold shift in animal studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects, 19-80 years of age;
* Confirmed diagnosis of advanced head and neck cancer or advanced lung cancer
* Voluntarily consent to participate in the study
* Females of childbearing potential should either be sexually inactive (abstinent) for 14 days prior to screening and throughout the study or be using one of the following acceptable birth control methods:
* IUD in place for at least 3 months prior to study;
* Barrier method (condom or diaphragm) with spermicide for at least 14 days prior to screening through study completion;
* Stable hormonal contraceptive for at least 3 months prior to study through completion of study;
* Surgical sterilization (vasectomy) of partner at least 6 months prior to study.
* Females of non-childbearing potential should be surgically sterile (bilateral tubal ligation with surgery at least 6 months prior to study, hysterectomy, or bilateral oophorectomy at least 2 months prior to study).

Exclusion Criteria:

* Subjects previously treated with chemotherapy, antibiotics, or diuretics known to cause hearing loss in the last 90 days
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, otologic, or psychiatric disease
* Presence of alcoholism or drug abuse
* Participation in another investigational drug or device clinical trial within 30 days prior to the study
* Female subjects who are pregnant or lactating

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-01-15 (Estimated); Primary Completion 2019-06-26 (Estimated); Study Completion 2019-09-23 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 12 months

SECONDARY OUTCOMES:
Reduction of hearing loss incidence and severity | From baseline through 1 month after last chemotherapy cycle
Reduction of tinnitus incidence and severity. | From baseline through 1 month after last chemotherapy cycle

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kil, MD, Study Director — Sound Pharmaceuticals, Inc.
Locations (1):
- VA Puget Sound Health Care, Seattle, Washington, United States

REFERENCES:
- [Background] Rybak LP, Whitworth C, Somani S. Application of antioxidants and other agents to prevent cisplatin ototoxicity. Laryngoscope. 1999 Nov;109(11):1740-4. doi: 10.1097/00005537-199911000-00003. PMID 10569399
- [Background] Rybak LP, Somani S. Ototoxicity. Amelioration by protective agents. Ann N Y Acad Sci. 1999 Nov 28;884:143-51. PMID 10842591
- [Background] Lynch ED, Gu R, Pierce C, Kil J. Reduction of acute cisplatin ototoxicity and nephrotoxicity in rats by oral administration of allopurinol and ebselen. Hear Res. 2005 Mar;201(1-2):81-9. doi: 10.1016/j.heares.2004.08.002. PMID 15721563
- [Background] Lynch ED, Gu R, Pierce C, Kil J. Combined oral delivery of ebselen and allopurinol reduces multiple cisplatin toxicities in rat breast and ovarian cancer models while enhancing anti-tumor activity. Anticancer Drugs. 2005 Jun;16(5):569-79. doi: 10.1097/00001813-200506000-00013. PMID 15846123
- [Background] Knight KR, Kraemer DF, Winter C, Neuwelt EA. Early changes in auditory function as a result of platinum chemotherapy: use of extended high-frequency audiometry and evoked distortion product otoacoustic emissions. J Clin Oncol. 2007 Apr 1;25(10):1190-5. doi: 10.1200/JCO.2006.07.9723. PMID 17401008
- [Background] Reavis KM, Phillips DS, Fausti SA, Gordon JS, Helt WJ, Wilmington D, Bratt GW, Konrad-Martin D. Factors affecting sensitivity of distortion-product otoacoustic emissions to ototoxic hearing loss. Ear Hear. 2008 Dec;29(6):875-93. doi: 10.1097/AUD.0b013e318181ad99. PMID 18753950
- [Background] Kim SJ, Park C, Han AL, Youn MJ, Lee JH, Kim Y, Kim ES, Kim HJ, Kim JK, Lee HK, Chung SY, So H, Park R. Ebselen attenuates cisplatin-induced ROS generation through Nrf2 activation in auditory cells. Hear Res. 2009 May;251(1-2):70-82. doi: 10.1016/j.heares.2009.03.003. Epub 2009 Mar 13. PMID 19286452
- [Background] Lynch E, Kil J. Development of Ebselen, a Glutathione Peroxidase Mimic, for the Prevention and Treatment of Noise-Induced Hearing Loss. Semin Hear 2009; 30(1): 047-055